CLINICAL TRIAL: NCT05667337
Title: Étude Clinique Ouverte et Prospective évaluant la sécurité et l'efficacité de la cornée biosynthétique CLP-PEG-MPC Chez Les Patients nécessitant Une kératoplastie Lamellaire antérieure Profonde à Haut Risque.
Brief Title: Open-label Prospective Clinical Trial Evaluating the Safety and Efficacy of Biosynthetic CLP-PEG-MPC Corneal Implants in Patients Undergoing High-risk Deep Anterior Lamellar Keratoplasty.
Acronym: CLP-PEG-MPC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: further biomaterial optimization
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20.017
Record Dates: First submitted 2020-10-06; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: High-risk Corneal Transplantation; Corneal Blindess; Corneal Inflammation; Deep Anterior Lamellar Keratoplasty
Keywords: cornea; biosynthetic implants; tissue regeneration
MeSH Terms: conditions — Keratitis; Corneal Diseases

STUDY DESIGN:
Intervention Model Description: Once qualified, subjects will be enrolled to receive a CLP-PEG-MPC implant by DALK. DALK surgery requires the precise dissection of the central 8 mm of the corneal stroma from the underlying posterior corneal layers (Dua layer, Descemet membrane and endothelium, approximately 30 microns thick). The dissection performed during DALK may perforate the posterior corneal layers, requiring conversion to full-thickness penetrating keratoplasty (PKP). Subjects who require conversion to PKP will receive a full-thickness human donor cornea as a safety measure and will be followed per protocol as a comparison group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLP-PEG-MPC DALK (Experimental): Subjects having successfully undergone implantation of CLP-PEG-MPC implant using DALK technique
  Interventions: Device: CLP-PEG-MPC
- HDC PKP (Active Comparator): Subjects having undergone DALK conversion to PKP using a human donor cornea tissue
  Interventions: Procedure: Human donor cornea penetrating keratoplasty

INTERVENTIONS:
Device: CLP-PEG-MPC — Implantation of a 500 um thick biosynthetic corneal implant utilizing DALK surgical technique
  Arms: CLP-PEG-MPC DALK
Procedure: Human donor cornea penetrating keratoplasty — Implantation of a human donor cornea graft utilizing PKP surgical technique
  Arms: HDC PKP

SUMMARY:
This is an open-label and prospective clinical trial, in which a maximum of 5 eyes of 5 patients will receive a CLP-PEG-MPC synthetic cornea during deep anterior lamellar keratoplasty (DALK) surgery and will be followed up over 24 months.

DETAILED DESCRIPTION:
This is a prospective open-label clinical trial of patients who will receive a CLP-PEG-MPC synthetic cornea during deep anterior lamellar keratoplasty (DALK) corneal transplantation surgery and be followed over 24 months. The primary objective is to demonstrate the safety and tolerability of CLP-PEG-MPC biosynthetic corneal implants. The secondary objective is to examine the preliminary efficacy of these implants to stimulate corneal tissue regeneration, provide optical clarity and improvement of vision. Randomization is not appropriate in a first-in-human pilot study. Blinding is not possible as surgeons can easily tell a cell-free implant apart from a donor allograft.

ELIGIBILITY:
Inclusion Criteria:

1. adult age (18 years or older at the time of subject eligibility visit)
2. able to provide signed, informed consent
3. unilateral corneal opacity not involving the posterior corneal layers (Descemet membrane and endothelium) for which DALK is indicated
4. visual acuity less than 20/200 in the affected eye and better than 20/50 in the contralateral eye (i.e. monocular blindness)
5. presence of at least one of the following high-risk criteria for corneal transplantation using a human cornea donor graft: 5i) inflammation 5ii) active infection 5iii) stromal neovascularization 5iv) neurotrophism 5v) autoimmune disease 5vi) previous DALK graft failure
6. availability for 24 months of postoperative follow-up

Exclusion Criteria:

1. Age under 18 years
2. Inability to give informed consent
3. Previous corneal perforation precluding DALK surgery
4. Endothelial pathology requiring penetrating keratoplasty
5. Limbal stem cell deficiency affection more than 50% of the limbus
6. Previous penetrating or endothelial keratoplasty
7. Bilateral blindness
8. Nystagmus
9. Uncontrolled glaucoma or intraocular pressure
10. Documented macular disease (age-relate macular degeneration, macula-involving retinal detachment, macular hole)
11. Documented amblyopia of surgical eye

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2040-01-01 (Estimated); Study Completion 2040-06-01 (Estimated)

PRIMARY OUTCOMES:
conjunctival inflammation | 24 months
  bulbar conjunctival inflammation (scale 0-none to 4-worse)
intraocular inflammation | 24 months
  anterior uveitis (SUN classification of cell and flare for anterior uveitis)
complications | 24 months
  occurence of implant-related complications
visual acuity - uncorrected | 24 months
  uncorrected visual acuity
visual acuity - best-spectacle correction | 24 months
  best-spectacle corrected visual acuity

SECONDARY OUTCOMES:
ocular pain | 24 months
  intensity of ocular pain and discomfort (questions 1,3, 10, 11 and 12 from Ocular Surface Disease Index questionnaire)
corneal thickness | 24 months
  central corneal pachymetry
corneal sensation | 24 months
  Central corneal esthesiometry using Cochet-Bonnet esthesiometer
Refraction | 24 months
  eye refractive error

IPD SHARING:
Plan to Share IPD: No